CLINICAL TRIAL: NCT07083141
Title: The Effect of Peer Mentoring on University Adjustment, Leadership Levels, and Professional Perception in Midwifery Students: A Randomized Controlled Trial
Brief Title: Peer Mentoring in Midwifery Students: Its Impact on University Adjustment, Leadership, and Professional Perception
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Suzi Özdemir, Assistant Professor, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Suzi-03
Record Dates: First submitted 2025-07-04; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Peer Mentorship; Peer Mentoring; Midwifery Education; MİDWİFERY STUDENT
Keywords: peer mentorship; peer mentoring; midwifery education; midwifery student

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mentor Intervention Group (Experimental)
  Interventions: Other: Peer Mentoring Program
- Mentor Control Group (No Intervention)
- Mentee Intervention Group (Experimental): Mentee Control Group
  Interventions: Other: Peer Mentoring Program
- Mentee Control Group (No Intervention)

INTERVENTIONS:
Other: Peer Mentoring Program — A 13-week peer mentoring program in which trained third-year midwifery students supported first-year students through regular meetings aimed at enhancing academic adaptation, confidence, and professional understanding.
  Arms: Mentee Intervention Group; Mentor Intervention Group

SUMMARY:
This study aimed to evaluate the effects of a peer mentoring program on first- and third-year midwifery students at a university in Türkiye. Peer mentoring involves experienced students (mentors) providing guidance and support to new students (mentees). A total of 120 students were randomly assigned to either a mentoring group or a control group. The program lasted for 13 weeks and included face-to-face meetings between mentors and mentees. The study was designed to assess how peer mentoring may contribute to students' university adjustment, leadership development, and perceptions of the midwifery profession.

DETAILED DESCRIPTION:
Starting university can be both exciting and overwhelming for students, particularly in health-related fields such as midwifery. Students often face challenges like adapting to academic demands, managing stress, and developing a professional identity. Peer mentoring is a supportive strategy in which more experienced students (mentors) help newcomers (mentees) by sharing their knowledge, experiences, and advice.

In this study, first- and third-year midwifery students at a university in Türkiye participated in a structured peer mentoring program. Third-year students were trained as mentors and paired with first-year mentees. Over the course of 13 weeks, mentors and mentees met regularly to discuss topics including academic concerns, campus life, and professional development.

The study was designed to examine the potential of peer mentoring as a support mechanism in midwifery education. The program aimed to help students adapt more effectively to university life, foster leadership skills among mentors, and support students' understanding and engagement with their future profession.

ELIGIBILITY:
Inclusion Criteria:

* Must be enrolled as a 1st-year or 3rd-year midwifery student at the university
* Must be attending classes regularly
* For mentors (3rd-year students): GPA must be 2.0 or higher
* Voluntary participation with signed informed consent

Exclusion Criteria:

* Having a diagnosed psychiatric condition
* Having communication disabilities
* Being on academic leave or not actively attending courses

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2025-07-02 (Actual)

PRIMARY OUTCOMES:
Change in University Adaptation Score After Peer Mentoring | Baseline and Week 13 (end of the semester)

SECONDARY OUTCOMES:
Change in Leadership Orientation Score Among Mentors | Baseline and Week 13 (end of the semester)
Change in Professional Perception Score Among Mentees | Baseline and Week 13 (end of the semester)

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University, Köseköy, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data (IPD) that underlie the results reported in this study (including anonymized survey responses and scale scores) will be shared.
  The data will be available beginning 6 months after publication of the main results, for researchers who provide a methodologically sound proposal.
  Data will be shared through institutional data-sharing agreements and will require ethics approval.
  Access will be granted for academic purposes only.